CLINICAL TRIAL: NCT00829322
Title: Modafinil for the Treatment of Fatigue in Lung Cancer: a Multicentre, Randomised, Double-blinded, Placebo-controlled Trial
Brief Title: Modafinil for the Treatment of Fatigue in Lung Cancer V9.0
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Modafinil/lung/09
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Experimental)
  Interventions: Drug: Modafinil
- Control group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Modafinil — Modafinil 100mg once daily for 14 days, increasing to 200mg once daily for a further 14 days
  Arms: Treatment group
Drug: Placebo — One capsule daily for 14 days, increasing to two capsules daily for 14 days
  Arms: Control group

SUMMARY:
Fatigue is a persistent, subjective sense of tiredness, which interferes with a person's usual ability to function. It is believed to be both the most common and the most distressing symptom experienced by those with cancer. Despite the magnitude of the problem, there has been inadequate research into the management of cancer-related fatigue.

Central nervous system (CNS) stimulants are the only class of drug established as being directly effective in relieving fatigue. Traditional stimulants, such as methylphenidate (Ritalin), can cause side-effects such as difficulty sleeping at night and anxiety. Modafinil is a relatively new stimulant with few side-effects. There is increasing evidence that modafinil can reduce fatigue in healthy individuals and patients with chronic, non-cancer conditions. No good quality studies have been published evaluating modafinil in patients with cancer, despite multiple calls for such research to be undertaken.

The investigators have completed a small study to determine the feasibility of undertaking a larger, high quality study to assess the effect of modafinil on fatigue in patients with lung cancer. Modafinil appeared to improve fatigue rapidly and was not associated with serious side-effects. Ten of the fifteen patients who completed the study chose to continue modafinil long-term. However, the study was too small for definite conclusions to be drawn.

This larger, definitive study, funded by a National Cancer Research Institute research award, will establish more clearly whether modafinil can improve fatigue in patients with lung cancer. Two hundred and six patients will be recruited from a number of sites across the UK. Half of the patients will take modafinil, and the other half will take a 'dummy' tablet every day for a month. The fatigue levels of the two groups will be compared. Confirmation that modafinil can relieve cancer-related fatigue could have a highly significant impact on the quality of life of the very large number of patients suffering from this common and distressing symptom.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Male or female, aged 18 years or above
* Diagnosed with NSCLC
* Stage 3a, 3b or stage 4 disease, or recurrent disease after surgery or radiotherapy
* WHO performance status of 0-2
* Participant has a screening score of 5 or more in a 10-point numerical rating scale (NRS) of fatigue severity within two weeks of enrolment
* Able (in the investigator's opinion) and willing to comply with all study requirements, including ability to participate for in study for 28 days
* Willing to allow his or her General Practitioner to be notified of participation in the study.

Exclusion Criteria:

* Received radiotherapy or chemotherapy within the last 4 weeks
* Commenced on an EGFR tyrosine kinase inhibitors eg Gefitinib and Erlotinib within the last 6 weeks.
* Commenced on antidepressants or steroids (corticosteroids and progestational steroids) within the last 2 weeks
* Received blood transfusion within the last 2 weeks
* Potentially fertile woman of child-bearing age
* Major anxiety requiring intervention in secondary care
* History of arrhythmia requiring medical intervention
* Uncontrolled hypertension with blood pressure greater than 160/100 mmHg
* History of cor pulmonale or left ventricular hypertrophy
* Currently taking warfarin
* Previous adverse reaction to modafinil or other CNS stimulant
* Scheduled elective surgery or other procedures requiring general anaesthesia during the study
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or affect the participant's ability to participate in the study
* Currently participating in another research study involving an investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2009-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
The fatigue subscale of the Functional Assessment of Chronic Illness Therapy measurement system | 28 days

SECONDARY OUTCOMES:
Epworth Sleepiness Scale | 28 days
Hospital Anxiety and Depression Scale | 28 days
Quality of life linear analogue scale | 28 days
Adverse events | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Bee Wee, PhD, Principal Investigator — University of Oxford
Locations (24):
- United Kingdom (24):
  - Stoke Mandeville Hospital, Aylesbury
  - Macclesfield District Hospital, Cheshire
  - University Hospital of North Tees, County Durham
  - Basildon and Thurrock University Hospitals, Essex
  - Basingstoke and North Hampshire Hospital, Hampshire
  - East Kent University Hospitals, Kent
  - Queen Elizabeth Hospital, Kings Lynn
  - University Hospital, Llandough
  - Royal Marsden Hospital Fulham Road, London
  - Royal Marsden Hospital Sutton, London
  - St George's Hospital, London
  - Christie Hospital, Manchester
  - Wythenshawe Hospital, Manchester
  - James Cook University Hospital, Middlesbrough
  - Harrogate and District NHS Foundation Trust, North Yorks
  - Churchill Hospital, Oxford
  - Papworth Hospital, Papworth Everard
  - Withybush General Hospital, Pembrokeshire
  - Peterborough District Hospital, Peterborough
  - Royal Surrey County Hospital, Surrey
  - Great Western Hospital, Swindon
  - Hillingdon Hospital, Uxbridge
  - Calderdale and Huddersfield NHS Foundation Trust, West Yorkshire
  - Mid Yorkshire Hospital NHS Trust, West Yorkshire

REFERENCES:
- [Derived] Spathis A, Fife K, Blackhall F, Dutton S, Bahadori R, Wharton R, O'Brien M, Stone P, Benepal T, Bates N, Wee B. Modafinil for the treatment of fatigue in lung cancer: results of a placebo-controlled, double-blind, randomized trial. J Clin Oncol. 2014 Jun 20;32(18):1882-8. doi: 10.1200/JCO.2013.54.4346. Epub 2014 Apr 28. PMID 24778393